CLINICAL TRIAL: NCT04692415
Title: The Differences Between Insulin Glargine U300 and Insulin Degludec U100 in Impact on the Glycaemic Variability, Oxidative Stress, Arterial Stiffness and the Lipid Profiles in Insulin naïve Patients Suffering From Type Two Diabetes Mellitus
Brief Title: Insulin Glargine U300 vs Insulin Degludec U100 in Impact on the Glycaemic and Cardiovascular Factors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Collaborators: Pavle Vrebalov Cindro (Unknown); Jonatan Vuković (Unknown); Darko Modun (Unknown); Božo Smajić (Unknown); Gordan Kardum (Unknown); Tina Tičinović Kurir (Unknown); Doris Rušić (Unknown); Ana Šešelja Perišin (Unknown); Josipa Bukić (Unknown)
Responsible Party: Principal Investigator, Mladen Krnic, Assistant professor, University of Split, School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 500-03/16-01/49
Record Dates: First submitted 2020-12-20; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus type 2; degludec; glargine U300; glucose variability; lipids; arterial stiffness; oxidative stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- degludec arm (Active Comparator): 25 patients were discontinued their previous therapy and given metformin alone (2 g/day) for seven days. After seven days they were randomized to first receive IDeg-100 In phase one they received IDeg-100 and metformin for 12 weeks. Phase one was followed by a second wash-up period in which patients received metformin alone again for seven days. In phase two, which also lasted for 12 weeks, patients were switched from IDeg-100 to IGlar-300 (and metformin was continued). The initial dose of both insulins was 0.2 IU/kg.
  Interventions: Drug: Degludec
- glargine arm (Active Comparator): 25 patients were discontinued their previous therapy and given metformin alone (2 g/day) for seven days. After seven days they were randomized to first receive IGlar-300 In phase one they received IGlar-300 and metformin for 12 weeks. Phase one was followed by a second wash-up period in which patients received metformin alone again for seven days. In phase two, which also lasted for 12 weeks, patients were switched from IGlar-300 to IDeg-100 (and metformin was continued). The initial dose of both insulins was 0.2 IU/kg.
  Interventions: Drug: Glargine U300

INTERVENTIONS:
Drug: Degludec — treatment of DM and it's affect on Glycaemic Variability, Oxidative Stress, Arterial Stiffness and the Lipid Profiles
  Arms: degludec arm
Drug: Glargine U300 — treatment of DM and it's affect on Glycaemic Variability, Oxidative Stress, Arterial Stiffness and the Lipid Profiles
  Arms: glargine arm

SUMMARY:
To compare the impact of insulin degludec (IDeg-100) and insulin glargine U300 (IGlar-300) on cardiovascular risk parameters - glycaemic variability (GV), oxidative stress, arterial stiffness and lipid parameters - in insulin naive patients with DMT2.

DETAILED DESCRIPTION:
We recruited a total of 25 patients (23 completed the study) with T2DM who had uncontrolled disease on two or more oral antidiabetic drugs. After the wash-up period, they were randomized alternately to first receive either IDeg-100 or IGlar-300 along with metformin. Each insulin was applied for 12 weeks. At the beginning and the end of each phase, biochemical and oxidative stress parameters were analysed and augmentation index was measured. On three consecutive days prior to each control point, patients performed a 7-point SMBG profile. Oxidative stress was assessed by measuring thiol groups and hydroperoxides (d-ROM) in serum. For augmentation index measuring, we used SphygmoCor (AtCor Medical, Sydney, Australia) which allow non-invasive measurement of AIx on radial artery using strain gauge transducer placed on the tip of a pencil-type tonometer. This method is based on the principle of applanation tonometry

ELIGIBILITY:
Inclusion Criteria:

* a history of DMT2 for at least 1 year
* aged between 18 and 65 years (women obligatory postmenopausal)
* uncontrolled glycaemia on two or more oral antidiabetic drugs
* no prior use of insulin
* HbA1c ≥7.5%
* receiving statins (if not on statins, they were put on it)
* not on antiaggregant therapy (if on antiaggregants, they were temporarily excluded from therapy)

Exclusion criteria:

* the presence of malignant disease
* chronic liver disease
* renal impairment with creatinine clearance < 60 ml/s
* severe cardiovascular disease or history of cardiovascular incidents (stroke, myocardial infarction, peripheral amputation)
* rheumatic and autoimmune diseases and the usage of glitazones or anticoagulant therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in glucose variability | 3 months
  Glucose variability will be assessed at the beginning and the end of each phase using 3-day 7-point SMBG and calculating coefficient of variation in % out of SMBG recordings
Changes from baseline in oxidative stress | 3 months
  Oxidative stress will be assessed at the beginning and the end of each phase by measuring thiol groups and hydroperoxides (d-ROM) in serum
Changes from baseline in arterial stiffness after treatment | 3 months
  Oxidative stress will be assessed at the beginning and the end of each phase by measuring augmentation index with SphygmoCor.

SECONDARY OUTCOMES:
Changes from baseline in total cholesterol | 3 months
  Total cholesterol concentration in mmol/L will be assessed at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in triglycerides | 3 months
  Triglyceride concentration in mmol/L will be assessed at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in LDL | 3 months
  Low density lipoprotein cholesterol concentration in mmol/L will be assessed at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in HDL | 3 months
  High density lipoprotein cholesterol concentration in mmol/L will be assessed at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in WBC | 3 months
  White blood count will be assessed at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in RBC | 3 months
  Red blood count will be assessed at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in platelets | 3 months
  Platelets count will be assessed at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in hemoglobin | 3 months
  Hemoglobin concentration in g/L will be assessed in at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in hematocrit | 3 months
  Hematocrit in L/L will be assessed in at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in MCV | 3 months
  Medium cellular volume in fL will be assessed in at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in liver enzymes | 3 months
  ALT, AST and GGT concentration in U/L will be assessed at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in LDH | 3 months
  Lactate dehydrogenase concentration in U/L will be assessed at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in ALP | 3 months
  Alkaline phosphatase concentration in U/L will be assessed at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit
Changes from baseline in CRP | 3 months
  C-reactive protein concentration in mg/L will be assessed at the beginning and the end of each phase by the automatic analyzer and enzymatic laboratory kit

CONTACTS AND LOCATIONS:
Locations (1):
- Klinički bolnički Centar Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: Yes
on request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: at any time
Access Criteria: health workers, health care organisations, health care providers, drug makers

REFERENCES:
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Eckel RH, Wassef M, Chait A, Sobel B, Barrett E, King G, Lopes-Virella M, Reusch J, Ruderman N, Steiner G, Vlassara H. Prevention Conference VI: Diabetes and Cardiovascular Disease: Writing Group II: pathogenesis of atherosclerosis in diabetes. Circulation. 2002 May 7;105(18):e138-43. doi: 10.1161/01.cir.0000013954.65303.c5. No abstract available. PMID 11994264
- [Background] Ceriello A, Esposito K, Piconi L, Ihnat MA, Thorpe JE, Testa R, Boemi M, Giugliano D. Oscillating glucose is more deleterious to endothelial function and oxidative stress than mean glucose in normal and type 2 diabetic patients. Diabetes. 2008 May;57(5):1349-54. doi: 10.2337/db08-0063. Epub 2008 Feb 25. PMID 18299315
- [Background] Monnier L, Colette C. Glycemic variability: should we and can we prevent it? Diabetes Care. 2008 Feb;31 Suppl 2:S150-4. doi: 10.2337/dc08-s241. PMID 18227477
- [Background] Monnier L, Mas E, Ginet C, Michel F, Villon L, Cristol JP, Colette C. Activation of oxidative stress by acute glucose fluctuations compared with sustained chronic hyperglycemia in patients with type 2 diabetes. JAMA. 2006 Apr 12;295(14):1681-7. doi: 10.1001/jama.295.14.1681. PMID 16609090
- [Background] Monnier L, Colette C, Owens DR. Glycemic variability: the third component of the dysglycemia in diabetes. Is it important? How to measure it? J Diabetes Sci Technol. 2008 Nov;2(6):1094-100. doi: 10.1177/193229680800200618. PMID 19885298
- [Background] Patoulias D, Papadopoulos C, Stavropoulos K, Zografou I, Doumas M, Karagiannis A. Prognostic value of arterial stiffness measurements in cardiovascular disease, diabetes, and its complications: The potential role of sodium-glucose co-transporter-2 inhibitors. J Clin Hypertens (Greenwich). 2020 Apr;22(4):562-571. doi: 10.1111/jch.13831. Epub 2020 Feb 14. PMID 32058679
- [Background] Vukovic J, Modun D, Budimir D, Sutlovic D, Salamunic I, Zaja I, Boban M. Acute, food-induced moderate elevation of plasma uric acid protects against hyperoxia-induced oxidative stress and increase in arterial stiffness in healthy humans. Atherosclerosis. 2009 Nov;207(1):255-60. doi: 10.1016/j.atherosclerosis.2009.04.012. Epub 2009 Apr 17. PMID 19457484
- [Background] Tamminen MK, Westerbacka J, Vehkavaara S, Yki-Jarvinen H. Insulin therapy improves insulin actions on glucose metabolism and aortic wave reflection in type 2 diabetic patients. Eur J Clin Invest. 2003 Oct;33(10):855-60. doi: 10.1046/j.1365-2362.2003.01220.x. PMID 14511356
- [Background] Gordin D, Saraheimo M, Tuomikangas J, Soro-Paavonen A, Forsblom C, Paavonen K, Steckel-Hamann B, Harjutsalo V, Nicolaou L, Pavo I, Koivisto V, Groop PH. Insulin exposure mitigates the increase of arterial stiffness in patients with type 2 diabetes and albuminuria: an exploratory analysis. Acta Diabetol. 2019 Nov;56(11):1169-1175. doi: 10.1007/s00592-019-01351-4. Epub 2019 May 22. PMID 31119456
- [Background] Aslan I, Kucuksayan E, Aslan M. Effect of insulin analog initiation therapy on LDL/HDL subfraction profile and HDL associated enzymes in type 2 diabetic patients. Lipids Health Dis. 2013 Apr 24;12:54. doi: 10.1186/1476-511X-12-54. PMID 23617853
- [Background] Home P, Bartley P, Russell-Jones D, Hanaire-Broutin H, Heeg JE, Abrams P, Landin-Olsson M, Hylleberg B, Lang H, Draeger E; Study to Evaluate the Administration of Detemir Insulin Efficacy, Safety and Suitability (STEADINESS) Study Group. Insulin detemir offers improved glycemic control compared with NPH insulin in people with type 1 diabetes: a randomized clinical trial. Diabetes Care. 2004 May;27(5):1081-7. doi: 10.2337/diacare.27.5.1081. PMID 15111525
- [Background] Heise T, Mathieu C. Impact of the mode of protraction of basal insulin therapies on their pharmacokinetic and pharmacodynamic properties and resulting clinical outcomes. Diabetes Obes Metab. 2017 Jan;19(1):3-12. doi: 10.1111/dom.12782. Epub 2016 Sep 26. PMID 27593206
- [Background] Tibaldi J, Hadley-Brown M, Liebl A, Haldrup S, Sandberg V, Wolden ML, Rodbard HW. A comparative effectiveness study of degludec and insulin glargine 300 U/mL in insulin-naive patients with type 2 diabetes. Diabetes Obes Metab. 2019 Apr;21(4):1001-1009. doi: 10.1111/dom.13616. Epub 2019 Jan 8. PMID 30552800
- [Background] Rosenstock J, Cheng A, Ritzel R, Bosnyak Z, Devisme C, Cali AMG, Sieber J, Stella P, Wang X, Frias JP, Roussel R, Bolli GB. More Similarities Than Differences Testing Insulin Glargine 300 Units/mL Versus Insulin Degludec 100 Units/mL in Insulin-Naive Type 2 Diabetes: The Randomized Head-to-Head BRIGHT Trial. Diabetes Care. 2018 Oct;41(10):2147-2154. doi: 10.2337/dc18-0559. Epub 2018 Aug 13. PMID 30104294
- [Derived] Vrebalov Cindro P, Krnic M, Modun D, Vukovic J, Ticinovic Kurir T, Kardum G, Rusic D, Seselja Perisin A, Bukic J. Comparison of the Impact of Insulin Degludec U100 and Insulin Glargine U300 on Glycemic Variability and Oxidative Stress in Insulin-Naive Patients With Type 2 Diabetes Mellitus: Pilot Study for a Randomized Trial. JMIR Form Res. 2022 Jul 8;6(7):e35655. doi: 10.2196/35655. PMID 35802405
- [Derived] Cindro PV, Krnic M, Modun D, Smajic B, Vukovic J. The differences between insulin glargine U300 and insulin degludec U100 in impact on the glycaemic variability, arterial stiffness and the lipid profiles in insulin naive patients suffering from type two diabetes mellitus - outcomes from cross-over open-label randomized trial. BMC Endocr Disord. 2021 Apr 29;21(1):86. doi: 10.1186/s12902-021-00746-1. PMID 33926446